CLINICAL TRIAL: NCT02788266
Title: Clinical Evaluation of Combined Surgical/ Restorative Treatment of Gingival Recession-type Defects Using Different Restorative Materials
Brief Title: Treatment of Gingival Recession-type Defects Using Different Restorative Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25901600-7587
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Gingival Recession; Tooth Abrasion
Keywords: Cervical lesion; gingival recession; restorative materials
MeSH Terms: conditions — Gingival Recession; Tooth Abrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- connective tissue graft+composite resin (Active Comparator): connective tissue graft plus composite resin
  Interventions: Procedure: connective tissue graft+composite resin
- connective tissue graft+ glass ionomer (Active Comparator): connective tissue graft plus resin modified glass ionomer cement
  Interventions: Procedure: connective tissue graft+ glass ionomer
- connective tissue graft+giomer (Active Comparator): connective tissue graft plus giomer
  Interventions: Procedure: connective tissue graft+giomer

INTERVENTIONS:
Procedure: connective tissue graft+composite resin — treatment of gingival recession associated with cervical lesions with sub epithelial connective tissue graft plus composite resin
  Arms: connective tissue graft+composite resin
Procedure: connective tissue graft+ glass ionomer — treatment of gingival recession associated with cervical lesions with sub epithelial connective tissue graft plus resin modified glass ionomer cement
  Arms: connective tissue graft+ glass ionomer
Procedure: connective tissue graft+giomer — treatment of gingival recession associated with cervical lesions with sub epithelial connective tissue graft plus giomer
  Arms: connective tissue graft+giomer

SUMMARY:
Background: The aim of this study was to evaluate the treatment of multiple gingival recessions associated with non-carious cervical lesions (NCCL) using a modified coronally advanced flap in combination with a sub-epithelial connective tissue graft (SCTG) on restored root surfaces.

Methods: Twenty-three systemically healthy subjects, who were positive for the presence of three cervical lesions associated with gingival recessions in three different adjacent teeth, were enrolled in the study. The NCCL were each restored prior to surgery by using one of three different materials: composite resin (group 1), resin-modified glass ionomer cement (group 2) or giomer (group 3). The defects were treated with SCTG. Clinical measurements, including plaque index (PI), bleeding on probing (BOP), relative recession height (rRH), probing depth (PD), cervical lesion height (CLH), relative clinical attachment level (rCAL), keratinized tissue height (KTH), keratinized tissue thickness (KTT), percentage of root coverage (RC), and percentage of cervical lesion height coverage (CLHC) were recorded at baseline, 3 and 6 months, and 1 year postoperatively.

DETAILED DESCRIPTION:
Gingival recession (GR) is defined as exposure of the root surface due to displacement of the gingival margin apical to the cemento-enamel junction (CEJ). Problems related to gingival recessions are dentin hypersensitivity, bacterial plaque accumulation, difficulty of maintaining oral health care and aesthetics, root caries and abrasions and fear of losing teeth6. Coronally advanced flap (CAF) is an effective periodontal plastic surgical procedure for the treatment of gingival recessions. The CAF with a subepithelial connective tissue graft (CAF+ SCTG) technique is reported as the gold standard and does enhance the probability of achieving complete root coverage.

Various dental materials and surgical approaches have been used to manage gingival recessions associated with cervical lesions for the most predictable combined surgical/restorative treatment.Restorative materials must be biocompatible to minimize their adverse effects on periodontal tissues induced by direct contact.Resin composites or resin modified glass ionomer cements have been commonly used to restore cervical lesions.Resin-ionomer materials have many properties such as biocompatibility with soft and hard tissues and displaying high marginal adaptation and minimal surface roughness as well as allowing them to be used successfully in the subgingival region. Composite resin materials have many advantages including aesthetics and surface characteristics in terms of finishing and polishing.

It has been reported that well-adapted and finished composite resins seem have no adverse effects on the periodontal margin. It has also been reported that the ageing of the composite resin restorations may produce gingival inflammation in subgingival areas. Fluoride-releasing resin materials with pre-reacted glass (PRG), called giomer, has been suggested to have good color matching, biocompatibility, smooth surface finish, fluoride release and fluoride recharge potential. It was reported in a randomized-controlled clinical trial that the use of CTG for treatment of root surfaces restored with giomer was effective over the 6-month period without any noxious effect on periodontal tissues.

Therefore, the aim of this study was to evaluate clinically the treatment of gingival recession associated with NCCL in resin modified glass ionomer cement (RMGI) or nano-filled resin composite (NRC) or giomer plus SCTG in the first year following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for the presence of three cervical lesions associated with multiple gingival recessions in three different adjacent teeth excluding molars;
2. Miller Class I gingival recession defect (≥2 and ≤5 mm) associated with buccal NCCL (lesion depth 1-2 mm);
3. Non-smoker;
4. Systemically and periodontally healthy;
5. Not taking medications known to interfere with periodontal tissue health or healing;
6. Probing depth (PD)≤3 mm;
7. Presence of ≥1 mm highly keratinized tissue apical to the root exposure, and presence of ≥0.8 mm-thick gingival tissue;
8. Absence of non-vital teeth, caries or restorations on cervical areas, severe occlusal interferences and previous surgery in the area.

Exclusion Criteria:

* inflammatory periodontal disease; previous surgical attempt to correct gingival recession; systemic disease or severe immune deficiency; coagulation defect or current anticoagulation treatment; addiction to drugs; inability or unwillingness to complete the trial; lack of linguistic skills; psychiatric disorders; refusal to sign the informed consent form; pregnancy; molar or premolar teeth with furcation involvement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
relative gingival recession height | one year post-op
  measured as distance from the most apical point of gingival margin to the incisional border of the tooth

SECONDARY OUTCOMES:
keratinized tissue width | one year
  measured from most apical point of the gingival margin to the mucogingival junction

CONTACTS AND LOCATIONS:
Overall Officials: gonen ozcan, Ph D, Study Director — Prof.dr.

IPD SHARING:
Plan to Share IPD: No